CLINICAL TRIAL: NCT00439153
Title: Quality of Surgical Field in Reconstructive Anterior Cruciate Ligament Surgery: Comparison of Tourniquet Cuff Pressure Determined by an Automated Limb Occlusion Pressure Measurement to a Standard Pressure of 300 mm Hg.
Brief Title: Minimizing Tourniquet Pressures in Paediatric Orthopaedic Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H06-03184
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Anterior Cruciate Ligament Repair

STUDY DESIGN:
Who Masked: Investigator

INTERVENTIONS:
Device: Tourniquet instrument capable of measuring LOP in combination with tourniquet cuffs — See Detailed Description.

SUMMARY:
Tourniquet cuffs are routinely used to stop blood flow in patients' arms or legs during surgery. This allows surgeons to better visualize anatomical structures during the procedure. Although complications after surgery are rare, patients sometimes suffer from pain or numbness in their limb and redness of the skin in the area where the cuff was applied. Using the lowest pressure possible minimizes the chance of these problems. Previous studies, conducted on adults, have shown that basing the cuff pressure on the minimum amount of pressure necessary to stop blood flow to the limb (known as limb occlusion pressure, or LOP) can lead to lower cuff pressures successfully being used. The goal of this study is to determine the magnitude by which tourniquet cuff pressure can be reduced in children using a tourniquet instrument capable of measuring LOP in combination with tourniquet cuffs selected to fit the size and contour of the limb. The tourniquet instrument and cuffs used in this study are all commercially available and approved for use with children.

Hypothesis:

It is hypothesized that use of a commercially available tourniquet instrument capable of calculating limb occlusion pressure in combination with tourniquet cuffs selected and applied according to a standardized procedure will produce surgical fields of equal or superior quality with significantly lower tourniquet cuff pressures.

DETAILED DESCRIPTION:
1. Purpose The risk of tourniquet-related injury increases with increasing tourniquet cuff pressure, therefore techniques intended to minimise tourniquet cuff pressures should be compared to current standard methods. A commercially available pneumatic tourniquet capable of measuring the pressure needed to occlude blood flow to a limb, known as limb occlusion pressure, combined with contoured tourniquet cuffs has been shown to significantly decrease necessary cuff pressures in adult patients. The magnitude of reduction in cuff pressure in a paediatric population has not yet been determined. Results of this study may decrease the standard tourniquet pressures used by paediatric orthopaedic surgeons, thereby reducing the risk of tourniquet-related injuries.
2. Justification Many studies have shown that both tourniquet pressure and time should be minimised to reduce the risk of tourniquet related injuries and post operative complaints. As the purpose of the tourniquet is to maintain a bloodless surgical field, in theory the minimum cuff pressure required to occlude arterial flow (the 'Limb Occlusion Pressure' or LOP), plus a safety margin to allow for changing conditions during the procedure, should be used. In practice, most surgeons use a standard pressure based on experience, or based on an indirect measurement of systolic blood pressure.

   Previous studies have shown that basing the cuff pressure on the LOP measured on each patient immediately prior to limb exsanguination and cuff inflation can lead to lower cuff pressures being used on many adult patients. This technique directly measures the cuff pressure required to occlude flow, thereby accounting for the individual patient's limb and vessel characteristics as well as the type and fit of the cuff. Unfortunately, the standard method of measuring limb occlusion pressure (monitoring a distal artery with a Doppler ultrasound probe while slowly increasing cuff pressure) is awkward and time consuming. A tourniquet device that allows automatic measurement of LOP at the start of each surgical procedure is now commercially available. This device has been shown to significantly reduce cuff inflation pressures necessary to occlude blood flow in adults; however, the magnitude of reduction in cuff pressure has not previously been determined in a paediatric population.

   Previous studies also suggest that wider tourniquet cuffs that are contoured such that they match the taper of the limb when applied occlude blood flow at lower pressures in adults. It is of interest to determine if wider cuffs, and contour cuffs designed to better fit tapered limbs, in combination with LOP calculation, allow for significantly lower cuff pressures in practical use on paediatric patients.
3. Objectives Quality of surgical field will be the primary outcome of this study. Secondary outcomes will include reduction in tourniquet cuff pressures and incidence of neurapraxias.
4. Research Method The target population will include subjects scheduled to receive anterior cruciate reconstruction at BC Children's Hospital by Dr. Chris Reilly. Subjects will prospectively be randomized into two groups. In the control group, tourniquet inflation pressures consistent with the current standard of care at BC Children Hospital will be used. In the experimental group, tourniquet inflation pressures will be determined by an automated calculation of limb occlusion pressure plus a predetermined safety margin. This technique has previously been shown to be equivalent to the Doppler technique for determining tourniquet inflation pressures, which is the gold standard. This is a non-inferiority trial with a power set at 0.8 and an alpha of 0.05. The estimated sample size is 21 patients in each group.
5. Method The study is a single blinded, randomised, prospective clinical comparison of two techniques used for determining tourniquet cuff pressure. The quality of surgical field will be compared in the experimental group (cuff pressure determined by LOP calculation) and the control group (standard cuff pressure of 300 mm Hg).

At the start of the study, 21 sealed envelopes indicating 'LOP + paediatric cuff' and 21 indicating 'standard pressure + standard cuff' will be prepared. The envelopes will be placed in blocks of 4 and 6 in order to minimise the predictive effect. After the grouping of the patient is determined, the person normally responsible for tourniquet cuff application will select an envelope and apply the indicated cuff at the indicated pressure.

For the 'LOP + paediatric cuff' group, cuff selection and application will be based on a standardized guide used to determine the most appropriate size and shape of cuff for the given limb. See cuff application guidelines (attached). Once the indicated cuff has been applied, the photoplethysmographic LOP sensor will be clipped to a toe of the affected leg, systolic blood pressure (SBP) will be recorded, and the automated LOP routine activated. LOP and recommended tourniquet pressure (RTP = LOP + predetermined margin) will be displayed within 1 minute and recorded. The limb will then be exsanguinated following the surgeon's usual procedure and the cuff inflated to the RTP.

For the 'standard pressure + standard cuff' group, cuff selection and application will be made based on the principal investigator's current practice. The limb will then be exsanguinated following the surgeon's usual procedure and the cuff inflated to a standard pressure, based on current practice and predetermined by the surgeon to be acceptable.

At the surgeon's discretion, the cuff pressure may be increased or decreased at any time during the procedure, with SBP, time, and the reason for change recorded. Immediately following the end of the procedure, the surgeon (principal investigator) will rate the overall quality of the surgical field using a visual analogue scale. He will also be provided with an area to comment on visualization capabilities during specific aspects of the procedure or any difficulties that may have occurred. Tourniquet inflation time and variation in SBP taken from the anaesthetists chart will be recorded. Incidence of post operative neurapraxias will also be determined.

Patient recruitment and enrolment will continue until enough subjects have been recruited to show statistical significance, which is currently estimated to be 21 subjects per group. Differences in the quality of the surgical field and tourniquet inflation pressures will be compared between the two groups, in addition to incidence of neurapraxias.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be selected from the primary investigator's patients scheduled for anterior cruciate ligament repair surgery

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Quality of surgical field

SECONDARY OUTCOMES:
Average tourniquet cuff pressure
Incidence of neurapraxias

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Reilly, MD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada